CLINICAL TRIAL: NCT06769178
Title: Effect of Virtual Reality-Based Interventions on Clinical and Neuroplasticity, Brain Functional Resting State Networks in Cerebral Palsy Rehabilitation
Brief Title: How Much Virtual Reality Intervention Improve the Balance of Patients with Cerebral Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SimayA
Record Dates: First submitted 2024-10-02; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy
Keywords: adult cerebral palsy; functional magnetic reasonance imaging; virtual reality; becure systems; balance; resting state functional magnetic reasonance imaging
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Serious Game Group (Experimental): BecureBalance and WesenseSystems will be used.Games'll be chosen to improve balance and empowerment,and game levels will be adjusted according to the condition of the participants.Balance Adventure is a game that involves transferring weight in 4 directions.At level 1,the goal is to reach the exit by collecting all the stars. At level 3,the goal is to collect stars on a moving surface and move the ball without dropping it.Balance Surf game is played with weight transfer from right to left and forward.The aim of the game is to earn points by steering the surfboard on the screen,collecting stars and gift wrap objects.Sizing Ball and Aerobat games are played by connecting a wearable sensor to the muscle group that the participants want to exercise.By calibrating this sensor, we can assume the angle we want is 0,and when more than the angle we set is made,movement will be revealed in the game.For this,lower extremity muscles will be exercised with these games by wearing a resistance band.
  Interventions: Other: Virtual Reality based
- Control Group (Other): Participants in the control group will receive a total of 16 sessions of structured NGT-based exercise applications prepared by the researchers.For this, involving balance and strengthening'll be applied, focusing mainly on lower extremity movements. For warm-up exercises, trunk rotation, shoulder rotation, hip rotation and toe-to-toe elevation and descent'll be performed for 10 minutes.Strengthening exercises'll mostly focus on the lower extremity muscles.These exercises'll be practiced for 20 minutes, and the participants'll be given the following exercises while the weight is tied. Each exercise'll be done in 2 sets of 10 repetitions.Balance exercises'll be practiced statically and dynamically for 20 minutes with 2 sets of 10 repetitions.
  Interventions: Other: Virtual Reality based

INTERVENTIONS:
Other: Virtual Reality based — Participants will receive treatment by a specialist physiotherapist for a total of 16 sessions, 2 days a week on non-consecutive days for 8 weeks. Both groups will receive neurodevelopmental treatment (NGT) for 16 sessions. While the control group will receive traditional balance training in each session, the VR group will play virtual reality-based games.
  Other Names: Neurodevelopmental based

SUMMARY:
The purpose of this clinical study is to investigate how effective virtual reality applications are in adult cerebral palsy rehabilitation.

The main questions it aims to answer are:

Do virtual reality interventions (of Becure Balance and Becure Wesense Systems) improve balance and is this improvement reflected in the clinic? Is there a change in brain functional resting state networks after virtual reality interventions?

ELIGIBILITY:
Inclusion Criteria:

Being diagnosed with unilateral spastic type cerebral palsy (hemiplegic type) / Being between the ages of 18-30 / Being able to walk independently (GMFCS I-II) / Not having Botox application in the last six months / Not using any medication that will affect the study process

Exclusion Criteria:

Having a history of epileptic attacks / Having >2 spasticity in any joint according to the modified Ashworth scale / Having severe depression according to the Beck Depression Inventory /Having hearing-vision problems

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength Assessment | up to 8 weeks
  Muscle strength is an important component of health. Muscle weakness is seen in the presence of neurologicaldiseases and therefore muscle strength measurement is important for general health assessment. The most common equipment or methods that provide quantitative measurements of strength, such as isokinetic and portable dynamometers, have been shown to provide valid and reliable measurements. The muscle strengths of the participants in the lower extremity (hip flexor, extensor, abductor and adductor, knee flexor and extensor, ankle dorsi-plantar flexor) muscle groups will be measured with a handheld dynamometer.
Timed Up and Go Test (TUG) | up to 8 weeks
  TUG is a rapid test used in clinic as an outcome measure to assess functional mobility as well as static and dynamic balance. It's based on the length of time which takes for an individual to get up from a chair, walk 3 meters at a comfortable (or fastest) pace, turn (or touch the wall), walk to chair and sit down again.
Berg Balance Scale (BBS) | up to 8 weeks
  The BBS, developed by Berg et al (1995) and used in the assessment of balance, is a four-point scale that rates patients' balance from easy to difficult (0: cannot do, 4: does independently). During the test consisting of 14 items, steps, rulers, stopwatches and chairs are used. The test evaluates postural control and fall risk. The maximum total score is 56 points. 0-20: high fall risk, 21-40: moderate fall risk, 41-56: low fall risk. The Turkish validity and reliability of the scale was made by Şahin et al (2008).

SECONDARY OUTCOMES:
fMRI scan | up to 8 weeks
  High-resolution (1 x 1 x 1 mm isotropic) sagittal 190 slices will be acquired with a T1-weighted imaging sequence (TR/TE: 7.7/3.7 ms;, FA: 8°; FOV: 256 x 256). Functional resting state data will be acquired with a single-shot echo planar imaging (EPI) sequence of 300 dynamic acquisitions consisting of 35 slices of 4 mm thickness (TR/TE: 2230/30 ms, FA: 77°; matrix: 80x80) and will last approximately 11 minutes. Magnetic field maps will be recorded in order to correct signal distortions caused by tissue inhomogeneities in the magnetic field during the analysis phase before functional acquisition. Participants will be asked to fix their gaze on a point by keeping their eyes open during functional acquisitions. Participants will be informed that they can close their eyes and rest during the other stages of the acquisitions. fMRI acquisitions will be completed in approximately 30 minutes, including the preparation stages. The MRI acquisition sequences will be as follows: Survey, Resting S

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] You SH, Jang SH, Kim YH, Kwon YH, Barrow I, Hallett M. Cortical reorganization induced by virtual reality therapy in a child with hemiparetic cerebral palsy. Dev Med Child Neurol. 2005 Sep;47(9):628-35. PMID 16138671
- [Background] Wimalasundera N, Stevenson VL. Cerebral palsy. Pract Neurol. 2016 Jun;16(3):184-94. doi: 10.1136/practneurol-2015-001184. Epub 2016 Feb 2. PMID 26837375
- [Background] Warnier N, Lambregts S, Port IV. Effect of Virtual Reality Therapy on Balance and Walking in Children with Cerebral Palsy: A Systematic Review. Dev Neurorehabil. 2020 Nov;23(8):502-518. doi: 10.1080/17518423.2019.1683907. Epub 2019 Nov 1. PMID 31674852
- [Background] Upadhyay J, Ansari MN, Samad A, Sayana A. Dysregulation of multiple signaling pathways: A possible cause of cerebral palsy. Exp Biol Med (Maywood). 2022 May;247(9):779-787. doi: 10.1177/15353702221081022. Epub 2022 Mar 7. PMID 35253451
- [Background] Reyes F, Niedzwecki C, Gaebler-Spira D. Technological Advancements in Cerebral Palsy Rehabilitation. Phys Med Rehabil Clin N Am. 2020 Feb;31(1):117-129. doi: 10.1016/j.pmr.2019.09.002. Epub 2019 Nov 6. PMID 31760985
- [Background] Reid LB, Pagnozzi AM, Fiori S, Boyd RN, Dowson N, Rose SE. Measuring neuroplasticity associated with cerebral palsy rehabilitation: An MRI based power analysis. Int J Dev Neurosci. 2017 May;58:17-25. doi: 10.1016/j.ijdevneu.2017.01.010. Epub 2017 Jan 24. PMID 28130065
- [Background] Papageorgiou E, De Beukelaer N, Simon-Martinez C, Mailleux L, Van Campenhout A, Desloovere K, Ortibus E. Structural Brain Lesions and Gait Pathology in Children With Spastic Cerebral Palsy. Front Hum Neurosci. 2020 Jul 9;14:275. doi: 10.3389/fnhum.2020.00275. eCollection 2020. PMID 32733223
- [Background] Papadelis C, Ahtam B, Feldman HA, AlHilani M, Tamilia E, Nimec D, Snyder B, Ellen Grant P, Im K. Altered White Matter Connectivity Associated with Intergyral Brain Disorganization in Hemiplegic Cerebral Palsy. Neuroscience. 2019 Feb 10;399:146-160. doi: 10.1016/j.neuroscience.2018.12.028. Epub 2018 Dec 26. PMID 30593919
- [Background] Jaatela J, Nurmi T, Vallinoja J, Maenpaa H, Sairanen V, Piitulainen H. Altered corpus callosum structure in adolescents with cerebral palsy: connection to gait and balance. Brain Struct Funct. 2023 Nov;228(8):1901-1915. doi: 10.1007/s00429-023-02692-1. Epub 2023 Aug 24. PMID 37615759
- [Background] Hawe RL, Sukal-Moulton T, Dewald JP. The effect of injury timing on white matter changes in the corpus callosum following unilateral brain injury. Neuroimage Clin. 2013 Aug 8;3:115-22. doi: 10.1016/j.nicl.2013.08.002. eCollection 2013. PMID 24179855
- [Background] Hajebrahimi F, Velioglu HA, Bayraktaroglu Z, Helvaci Yilmaz N, Hanoglu L. Clinical evaluation and resting state fMRI analysis of virtual reality based training in Parkinson's disease through a randomized controlled trial. Sci Rep. 2022 May 16;12(1):8024. doi: 10.1038/s41598-022-12061-3. PMID 35577874
- [Background] Hadzagic-Catibusic F, Avdagic E, Zubcevic S, Uzicanin S. Brain Lesions in Children with Unilateral Spastic Cerebral Palsy. Med Arch. 2017 Feb;71(1):7-11. doi: 10.5455/medarh.2017.71.7-11. Epub 2017 Feb 5. PMID 28428665
- [Background] Erten AB, Tarakci D, Cacan MA. The Effectiveness of Video-Based Game Exercise Therapy Applications in Pes Planus Rehabilitation: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Sep 11;12:e51772. doi: 10.2196/51772. PMID 37695657
- [Background] Coskun B, Ay S, Erol Barkana D, Bostanci H, Uzun I, Oktay AB, Tuncel B, Tarakci D. A physiological signal database of children with different special needs for stress recognition. Sci Data. 2023 Jun 14;10(1):382. doi: 10.1038/s41597-023-02272-2. PMID 37316526